CLINICAL TRIAL: NCT01244984
Title: A Long-term Study to Evaluate the Safety and Tolerability of Fluticasone Furoate (FF)/GW642444 Inhalation Powder and FF Inhalation Powder in Japanese Subjects With Asthma
Brief Title: A Long-term Safety Study of Fluticasone Furoate (FF)/GW642444 and FF in Japanese Subjects With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 113989
Record Dates: First submitted 2010-11-18; First posted 2010-11-22 (Estimated); Results first posted 2013-08-09 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: asthma; Fluticasone furoate; GW642444
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone Furoate/GW642444 (Experimental): Combination inhaled corticosteroid and long-acting beta2-agonist
  Interventions: Drug: Fluticasone Furoate/GW642444 Inhalation Powder
- Fluticasone Furoate (Experimental): Inhaled corticosteroid
  Interventions: Drug: Fluticasone Furoate Inhalation Powder

INTERVENTIONS:
Drug: Fluticasone Furoate/GW642444 Inhalation Powder — Fluticasone Furoate/GW642444 inhalation powder inhaled orally once daily for 52 weeks
  Arms: Fluticasone Furoate/GW642444
Drug: Fluticasone Furoate Inhalation Powder — Fluticasone Furoate inhalation powder inhaled orally once daily for 52 weeks
  Arms: Fluticasone Furoate

SUMMARY:
The primary purpose of the study is to assess the safety and tolerability of 52-week teatment with fluticasone furoate/GW642444 inhalation powder once-daily and FF inhalation powder once-daily in Japanese adult subjects with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Out patient at least 18 years of age
* Both genderds; females of childbearing potential must be willing to use birth control method
* A diagnosis of asthma at least 6 months prior to Screening
* A best FEV1 of at least 50% of the predicted nomal value at Screening
* Subjects have been receiving maintanance therapy for asthma, for at least 4 weeks prior to Screening

Exclusion Criteria:

* History of life-threating asthma
* Respiratory infection or oral candidiasis
* Asthma exacerbation within 12 weeks
* Concurrent respiratory disease or other disease that would confound study participation or affect subject safety
* Allergies to study drugs, study drugs7 excipients, medications related to study drugs
* Taking another investigational medication or medication prohibited for use during this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2010-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- Japan (15):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Toyama

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- [Derived] O'Byrne PM, Jacques L, Goldfrad C, Kwon N, Perrio M, Yates LJ, Busse WW. Integrated safety and efficacy analysis of once-daily fluticasone furoate for the treatment of asthma. Respir Res. 2016 Nov 24;17(1):157. doi: 10.1186/s12931-016-0473-x. PMID 27881132
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 113989 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113989 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113989 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113989 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113989 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113989 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113989 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following screening (Visit1) and a 2-week Run-in Period during which participants continued to use their respective asthma therapy at a fixed dose. Participants who met continuation criteria at the end of Run-in Period (Visit 2) were allocated to a 52-Week Treatment Period.
Groups:
- FF/GW642444 100/25 µg: Participants received Fluticasone Furoate (FF)/GW642444 inhalation powder 100/25 micrograms (µg ) once daily (OD) in the evening from the Dry Powder Inhalator (DPI) over the 52 week treatment period.
- FF/GW642444 200/25 µg: Participants received FF/GW642444 inhalation powder 200/25 µg OD in the evening from the DPI over the 52 week treatment period.
- FF 100 µg: Participants received FF inhalation powder 100 µg OD in the evening from the the DPI over the 52 week treatment period.
Period: Overall Study
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Started | 60 | 93 | 90
Completed | 55 | 79 | 86
Not Completed | 5 | 14 | 4
Not completed — Adverse Event | 2 | 11 | 2
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Protocol Defined Stopping Criteria | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- FF/GW642444 100/25 µg: Participants received Fluticasone Furoate (FF)/GW642444 inhalation powder 100/25 micrograms (µg) once daily (OD) in the evening from the Dry Powder Inhalator (DPI) over the 52 week treatment period.
- Total: Total of all reporting groups
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg | Total
Number analyzed (Participants) | 60 | 93 | 90 | 243
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.3 (13.74) | 52.6 (15.05) | 46.8 (15.46) | 50.1 (15.06)
Gender [Count of Participants; unit: Participants]
  Female | 38 | 49 | 54 | 141
  Male | 22 | 44 | 36 | 102
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Japanese Heritage | 60 | 93 | 90 | 243

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Non-serious Adverse Event (AE) and Any Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, may jeopardize the participant or require medical or surgical intervention to prevent one of the other outcomes listed in the definition above, or is an event of possible drug-induced liver injury. Refer to the general AE/SAE module for a list of AEs (occurring at a frequency threshold >=5%) and SAE.
Time Frame: From the start of investigational product to the last dose of treatment (up to Week 52/Withdrawal [WD])
Population: Intent-to-Treat (ITT) Population: all participants who had been randomized to and received at least one dose of randomized medication in the treatment period
Measure: Number; unit: Participants
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Number analyzed (Participants) | 60 | 93 | 90
Participants
  Any SAE | 4 | 7 | 1
  Any Non-serious AE | 52 | 77 | 72

2. Secondary Outcome: Laboratory Parameters of Basophils, Eosinophils, Lymphocytes, Monocytes, and Total Neutrophils at Baseline (Week -2), Week 12, Week 24, and Week 52/WD
Description: Blood samples were collected for measurement at the following scheduled time points: Baseline (Week -2), Week 12, Week 24 and Week 52/WD.
Time Frame: Baseline (Week -2), Week 12, Week 24, and Week 52/WD
Population: ITT Population. Only participants remaining in the study and contributing evaluable data at the indicated time points were analyzed.; thus the number of participants analyzed reflects everyone in the ITT Population. The number of participants assessed for each parameter is indicated by "n=X, X".
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Number analyzed (Participants) | 60 | 93 | 90
Percentage
  Basophils, Baseline, n=60,93,90 | 0.78 (0.509) | 0.71 (0.419) | 0.79 (0.508)
  Basophils, Week 12, n=58, 90, 87 | 0.76 (0.473) | 0.67 (0.414) | 0.79 (0.542)
  Basophils, Week 24, n=58, 83, 86 | 0.74 (0.510) | 0.66 (0.392) | 0.72 (0.408)
  Basophils, Week 52/WD, n=60, 90, 89 | 0.77 (0.510) | 0.64 (0.383) | 0.72 (0.482)
  Eosinophils, Baseline, n=60,93,90 | 5.59 (4.476) | 5.03 (3.843) | 5.32 (3.167)
  Eosinophils, Week 12, n=58, 90, 87 | 5.22 (3.257) | 4.01 (3.112) | 4.90 (3.496)
  Eosinophils, Week 24, n=58, 83, 86 | 4.88 (3.678) | 4.00 (2.753) | 4.37 (3.061)
  Eosinophils, Week 52/WD, n=60, 90, 89 | 4.89 (3.981) | 4.27 (3.247) | 4.60 (3.090)
  Lymphocytes, Baseline, n=60, 93, 90 | 30.49 (5.948) | 30.95 (7.504) | 31.26 (6.150)
  Lymphocytes, Week 12, n=58, 90, 87 | 29.22 (6.891) | 29.15 (6.378) | 29.35 (7.274)
  Lymphocytes , Week 24, n=58, 83, 86 | 29.06 (6.269) | 28.40 (6.282) | 28.83 (6.343)
  Lymphocytes, Week 52/WD, n=60, 90, 89 | 30.01 (6.702) | 27.67 (7.913) | 29.04 (7.047)
  Monocytes, Baseline, n=60,93,90 | 5.23 (1.307) | 5.39 (1.408) | 5.35 (1.442)
  Monocytes, Week 12, n=58, 90, 87 | 5.65 (1.187) | 5.61 (1.626) | 5.65 (1.639)
  Monocytes, Week 24, n=58, 83, 86 | 5.51 (1.571) | 5.52 (1.321) | 5.41 (1.370)
  Monocytes, Week 52/WD, n=60, 90, 89 | 5.59 (1.637) | 5.72 (1.366) | 5.59 (1.516)
  Total neutrophils, Baseline, n=60,93,90 | 57.91 (8.064) | 57.92 (8.103) | 57.28 (7.467)
  Total neutrophils, Week 12, n=58, 90, 87 | 59.14 (7.785) | 60.57 (7.474) | 59.31 (8.642)
  Total neutrophils, Week 24, n=58, 83, 86 | 59.82 (7.893) | 61.37 (6.790) | 60.64 (7.358)
  Total neutrophils, Week 52/WD, n=60, 90, 89 | 58.54 (8.910) | 61.70 (8.326) | 60.05 (7.883)

3. Secondary Outcome: Laboratory Parameters of Eosinophils, Platelet Count, White Blood Cell (WBC), and Total Neutrophils at Baseline (Week -2), Week 12, Week 24, and Week 52/WD
Description: as for outcome 2
Time Frame: Baseline (Week -2), Week 12, Week 24, and Week 52/WD
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 per liter (Gi/L)
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Number analyzed (Participants) | 60 | 93 | 90
10^9 per liter (Gi/L)
  Eosinophils, Baseline, n=60, 93, 90 | 0.338 (0.2514) | 0.323 (0.2591) | 0.323 (0.2042)
  Eosinophils, Week 12, n=58, 90, 87 | 0.306 (0.2106) | 0.245 (0.2057) | 0.286 (0.2154)
  Eosinophils, Week 24, n=58, 83, 86 | 0.282 (0.2244) | 0.247 (0.1864) | 0.256 (0.1907)
  Eosinophils, Week 52/WD, n=60, 90, 89 | 0.290 (0.2399) | 0.281 (0.2332) | 0.285 (0.2032)
  Platelet count, Baseline, n=60, 93, 90 | 252.4 (53.41) | 257.1 (64.98) | 254.1 (60.77)
  Platelet count, Week 12, n=58, 90, 87 | 263.9 (62.25) | 269.3 (60.55) | 259.0 (54.00)
  Platelet count, Week 24, n=58, 83, 86 | 261.1 (62.25) | 270.2 (66.60) | 260.1 (58.84)
  Platelet count, Week 52/WD, n=60, 90, 89 | 267.2 (54.93) | 276.7 (68.64) | 270.3 (63.75)
  WBC, Baseline, n=60, 93, 90 | 6.24 (1.716) | 6.39 (1.503) | 6.13 (1.495)
  WBC, Week 12, n=58, 90, 87 | 5.90 (1.642) | 6.11 (1.462) | 5.95 (1.636)
  WBC, Week 24, n=58, 83, 86 | 5.86 (1.541) | 6.19 (1.743) | 6.01 (1.564)
  WBC, Week 52/WD, n=60, 90, 89 | 6.11 (1.625) | 6.45 (1.530) | 6.24 (1.511)
  Total neutrophils, Baseline, n=60, 93, 90 | 3.661 (1.3444) | 3.734 (1.2446) | 3.536 (1.1080)
  Total neutrophils, Week 12, n=58, 90, 87 | 3.522 (1.2140) | 3.729 (1.1131) | 3.567 (1.2419)
  Total neutrophils, Week 24, n=58, 83, 86 | 3.522 (1.1186) | 3.833 (1.2812) | 3.690 (1.2837)
  Total neutrophils, Week 52/WD, n=60, 90, 89 | 3.585 (1.2570) | 4.010 (1.2422) | 3.795 (1.2221)

4. Secondary Outcome: Laboratory Parameter of Hemoglobin at Baseline (Week -2), Week 12,Week 24, and Week 52/WD
Description: as for outcome 2
Time Frame: Baseline (Week -2), Week 12, Week 24, and Week 52/WD
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Number analyzed (Participants) | 60 | 93 | 90
Grams per liter (g/L)
  Baseline, n=60, 93, 90 | 135.7 (15.88) | 141.1 (16.34) | 138.6 (15.61)
  Week 12, n=58, 90, 87 | 138.2 (15.10) | 140.6 (15.58) | 139.1 (14.47)
  Week 24, n=58, 83, 86 | 137.4 (15.45) | 140.8 (15.99) | 139.0 (14.92)
  Week 52/WD, n=60, 90, 89 | 136.4 (14.16) | 139.0 (15.91) | 136.7 (15.62)

5. Secondary Outcome: Laboratory Parameter of Hematocrit at Baseline (Week -2), Week 12, Week 24, and Week 52/WD
Description: as for outcome 2
Time Frame: Baseline (Week -2), Week 12, Week 24, and Week 52/WD
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Proportions of I
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Number analyzed (Participants) | 60 | 93 | 90
Proportions of I
  Baseline, n=60, 93, 90 | 0.4214 (0.04429) | 0.4374 (0.04417) | 0.4319 (0.04090)
  Week 12, n=58, 90, 87 | 0.4288 (0.04224) | 0.4325 (0.04199) | 0.4283 (0.03870)
  Week 24, n=58, 83, 86 | 0.4238 (0.04228) | 0.4333 (0.04277) | 0.4288 (0.03858)
  Week 52/WD, n=60, 90, 89 | 0.4194 (0.03921) | 0.4272 (0.04367) | 0.4215 (0.04138)

6. Secondary Outcome: Laboratory Parameter of Red Blood Cell Count at Baseline (Week -2), Week 12, Week 24, and Week 52/WD
Description: as for outcome 2
Time Frame: Baseline (Week -2), Week 12, Week 24, and Week 52/WD
Population: ITT Population. Only participants remaining in the study and contributing evaluable data at the indicated time points were analyzed; thus the number of participants analyzed reflects everyone in the ITT Population. The number of participants assessed for each parameter is indicated by "n=X, X".
Measure: Mean (Standard Deviation); unit: 10^12 per liter (Ti/L)
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Number analyzed (Participants) | 60 | 93 | 90
10^12 per liter (Ti/L)
  Baseline, n=60, 93, 90 | 4.557 (0.4987) | 4.714 (0.4804) | 4.689 (0.4493)
  Week 12, n=58, 90, 87 | 4.656 (0.4540) | 4.685 (0.4888) | 4.696 (0.4267)
  Week 24, n=58, 83, 86 | 4.626 (0.4679) | 4.687 (0.4898) | 4.681 (0.4357)
  Week 52/WD, n=60, 90, 89 | 4.603 (0.4469) | 4.671 (0.5082) | 4.664 (0.4643)

7. Secondary Outcome: Laboratory Parameter of Albumin and Total Protein (TP) at Baseline (Week -2), Week 12, Week 24, and Week 52/WD
Description: as for outcome 2
Time Frame: Baseline (Week -2), Week 12, Week 24, and Week 52/WD
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Number analyzed (Participants) | 60 | 93 | 90
g/L
  Albumin, Baseline, n=60, 93, 90 | 44.3 (2.72) | 44.8 (2.59) | 44.7 (2.86)
  Albumin, Week 12, n=58, 90, 87 | 44.3 (2.37) | 44.1 (2.66) | 44.3 (2.69)
  Albumin, Week 24, n=58, 83, 86 | 43.6 (2.52) | 43.9 (2.67) | 43.7 (2.69)
  Albumin, Week 52/WD, n=60, 90, 89 | 43.5 (2.49) | 43.4 (3.03) | 43.8 (2.72)
  TP, Baseline, n=60, 93, 90 | 73.3 (4.36) | 73.6 (3.62) | 74.6 (4.08)
  TP, Week 12, n=58, 90, 87 | 73.8 (3.70) | 73.0 (3.83) | 74.4 (4.56)
  TP, Week 24, n=58, 83, 86 | 72.3 (4.49) | 72.4 (3.92) | 73.3 (3.78)
  TP, Week 52/WD, n=60, 90, 89 | 71.5 (3.55) | 71.4 (3.60) | 72.5 (4.15)

8. Secondary Outcome: Laboratory Parameter of Alkaline Phosphatase (AP), Alanine Amino Transferase (ALT), Aspartate Amino Transferase (AST), Creatine Kinase, Gamma Glutamyl Transferase (GGT), and Lactate Dehydrogenase (LDH) at BL (Week -2), Week 12, Week 24, and Week 52/WD
Description: Blood samples were collected for measurement at the following scheduled time points: Baseline (BL) (Week -2), Week 12, Week 24 and Week 52/WD.
Time Frame: Baseline (Week -2), Week 12, Week 24, and Week 52/WD
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: International unit per liter (IU/L)
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Number analyzed (Participants) | 60 | 93 | 90
International unit per liter (IU/L)
  AP, Baseline, n=60, 93, 90 | 209.9 (57.34) | 222.7 (62.97) | 217.1 (64.13)
  AP, Week 12, n=58, 90, 87 | 217.9 (56.39) | 214.9 (56.73) | 220.3 (59.92)
  AP, Week 24, n=58, 83, 86 | 212.3 (59.48) | 216.4 (57.33) | 215.9 (58.96)
  AP, Week 52/WD, n=60, 90, 89 | 223.1 (64.76) | 219.9 (60.27) | 217.0 (57.89)
  ALT, Baseline, n=60, 93, 90 | 19.0 (9.69) | 22.3 (14.46) | 21.9 (16.43)
  ALT, Week 12, n=58, 90, 87 | 24.1 (23.12) | 21.3 (11.39) | 20.7 (11.44)
  ALT, Week 24, n=58, 83, 86 | 19.0 (11.52) | 20.7 (10.45) | 20.1 (10.35)
  ALT, Week 52/WD, n=60, 90, 89 | 21.8 (12.46) | 23.2 (13.52) | 23.0 (14.11)
  AST, Baseline, n=60, 93, 90 | 20.0 (5.48) | 22.0 (7.50) | 21.5 (8.99)
  AST, Week 12, n=58, 90, 87 | 23.2 (10.08) | 22.0 (7.59) | 21.7 (6.90)
  AST, Week 24, n=58, 83, 86 | 20.1 (5.72) | 21.2 (7.29) | 20.6 (6.02)
  AST, Week 52/WD, n=60, 90, 89 | 23.5 (9.47) | 23.3 (7.53) | 22.8 (6.75)
  Creatine Kinase, Baseline, n=60, 93, 90 | 111.9 (56.95) | 149.8 (134.73) | 104.0 (45.88)
  Creatine Kinase, Week 12, n=58, 90, 87 | 118.9 (84.32) | 134.0 (114.92) | 97.4 (39.32)
  Creatine Kinase, Week 24, n=58, 83, 86 | 115.4 (77.09) | 131.9 (118.86) | 103.0 (58.40)
  Creatine Kinase, Week 52/WD, n=60, 90, 89 | 105.3 (48.78) | 126.6 (105.24) | 99.9 (48.96)
  GGT, Baseline, n=60, 93, 90 | 25.4 (14.04) | 34.9 (42.70) | 30.0 (28.96)
  GGT, Week 12, n=58, 90, 87 | 28.1 (15.29) | 31.0 (32.21) | 28.2 (24.60)
  GGT, Week 24, n=58, 83, 86 | 24.7 (14.73) | 30.8 (39.66) | 26.5 (22.28)
  GGT, Week 52/WD, n=60, 90, 89 | 28.2 (16.85) | 34.6 (48.03) | 28.9 (24.59)
  LDH, Baseline, n=60, 93, 90 | 176.7 (23.78) | 186.9 (34.40) | 175.3 (27.97)
  LDH, Week 12, n=58, 90, 87 | 180.8 (32.66) | 185.7 (37.83) | 175.1 (28.03)
  LDH, Week 24, n=58, 83, 86 | 175.3 (29.35) | 184.4 (36.45) | 174.3 (27.84)
  LDH, Week 52/WD, n=60, 90, 89 | 179.5 (31.50) | 188.1 (39.96) | 177.9 (29.66)

9. Secondary Outcome: Laboratory Parameter of Bilirubin (Direct [BD], Indirect [BI], Total [BT], Creatinine, and Uric Acid at Baseline (Week -2), Week 12, Week 24, and Week 52/WD
Description: as for outcome 2
Time Frame: Baseline (Week -2), Week 12, Week 24, and Week 52/WD
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micromoles per Liter (µmol/L)
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Number analyzed (Participants) | 60 | 93 | 90
Micromoles per Liter (µmol/L)
  direct [BD], Baseline, n=60, 93, 90 | 3.220 (1.4459) | 3.236 (1.5838) | 3.401 (1.7851)
  direct [BD], Week 12, n=58, 90, 87 | 2.948 (1.2729) | 3.230 (1.5475) | 3.125 (1.6535)
  direct [BD], Week 24, n=58, 83, 86 | 3.214 (1.5717) | 3.338 (1.8484) | 2.903 (1.5970)
  direct [BD], Week 52/WD, n=60, 90, 89 | 2.850 (1.2057) | 3.344 (1.5574) | 3.055 (1.5569)
  indirect [BI], Baseline, n=60, 93, 90 | 7.495 (2.9883) | 7.079 (3.3788) | 7.125 (2.8688)
  indirect [BI], Week 12, n=58, 90, 87 | 7.017 (3.1004) | 7.600 (3.2131) | 6.938 (3.0451)
  indirect [BI], Week 24, n=58, 83, 86 | 7.842 (5.1553) | 7.747 (3.7420) | 6.760 (3.2222)
  indirect [BI], Week 52/WD, n=60, 90, 89 | 6.640 (2.7100) | 7.505 (3.5676) | 6.936 (3.4525)
  total [BT], Baseline, n=60, 93, 90 | 10.716 (4.1989) | 10.315 (4.7735) | 10.526 (4.3571)
  total [BT], Week 12, n=58, 90, 87 | 9.965 (4.1781) | 10.830 (4.5424) | 10.063 (4.3902)
  total [BT], Week 24, n=58, 83, 86 | 11.056 (6.4954) | 11.084 (5.4427) | 9.663 (4.4958)
  total [BT], Week 52/WD, n=60, 90, 89 | 9.491 (3.6503) | 10.849 (4.8513) | 9.991 (4.7177)
  Creatinine, Baseline, n=60, 93, 90 | 61.8800 (13.37091) | 66.4806 (15.94483) | 62.0568 (12.65536)
  Creatinine, Week 12, n=58, 90, 87 | 59.3042 (13.92743) | 62.9408 (15.71444) | 60.1628 (13.02866)
  Creatinine, Week 24, n=58, 83, 86 | 59.7614 (12.91371) | 64.5213 (15.90631) | 60.6773 (13.02242)
  Creatinine, Week 52/WD, n=60, 90, 89 | 60.4067 (12.52458) | 64.6204 (16.01762) | 61.3536 (14.38660)
  Uric acid, Baseline, n=60, 93, 90 | 304.0419 (90.67062) | 305.7784 (78.88104) | 310.6178 (96.11471)
  Uric acid, Week 12, n=58, 90, 87 | 302.6301 (86.10161) | 301.6297 (74.72395) | 303.8266 (87.04586)
  Uric acid, Week 24, n=58, 83, 86 | 299.6561 (78.45023) | 310.8726 (86.38513) | 308.5352 (91.73313)
  Uric acid, Week 52/WD, n=60, 90, 89 | 305.2315 (78.61596) | 300.3079 (82.30325) | 308.0262 (92.43123)

10. Secondary Outcome: Laboratory Parameter of Chloride, Carbon Dioxide Content/Bicarbonate, Glucose, Potassium, Sodium, and Urea/Blood Urea Nitrogen (BUN) at Baseline (Week -2), Week 12, Week 24, and Week 52/WD
Description: as for outcome 2
Time Frame: Baseline (Week -2), Week 12, Week 24, and Week 52/WD
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per Liter (mmol/L)
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Number analyzed (Participants) | 60 | 93 | 90
Millimoles per Liter (mmol/L)
  Chloride, BL, n=60, 93, 90 | 104.3 (1.97) | 104.2 (1.85) | 103.6 (1.60)
  Chloride, Week 12, n=58, 90, 87 | 105.9 (2.05) | 105.6 (2.38) | 105.6 (2.14)
  Chloride, Week 24, n=58, 83, 86 | 105.4 (2.04) | 105.0 (2.44) | 105.0 (2.16)
  Chloride, Week 52/WD, n=60, 90, 89 | 105.6 (2.19) | 105.3 (2.41) | 104.8 (2.12)
  CO2 content/Bicarbonate, BL, n=60, 93, 90 | 25.3 (2.02) | 25.0 (1.84) | 25.2 (1.95)
  CO2 content/Bicarbonate, Week 12, n=58, 90, 87 | 24.9 (2.01) | 24.8 (2.13) | 25.4 (1.81)
  CO2 content/Bicarbonate, Week 24, n=58, 83, 86 | 25.4 (2.26) | 25.3 (2.33) | 24.8 (2.32)
  CO2 content/Bicarbonate, Week 52/WD, n=60, 90, 88 | 24.9 (2.03) | 25.3 (2.14) | 25.1 (2.04)
  Glucose, BL, n=60, 93, 90 | 5.6685 (0.88699) | 5.7826 (0.98753) | 5.7669 (1.03176)
  Glucose, Week 12, n=58, 90, 87 | 5.5606 (1.07679) | 5.7848 (1.01409) | 5.7647 (1.05233)
  Glucose, Week 24, n=58, 83, 86 | 5.8228 (1.41235) | 5.8593 (0.97613) | 5.8169 (1.43353)
  Glucose, Week 52/WD, n=60, 90, 89 | 5.4455 (1.05905) | 5.7743 (1.00636) | 5.8572 (1.17153)
  Potassium, BL, n=60, 93, 90 | 4.04 (0.279) | 4.13 (0.332) | 4.12 (0.338)
  Potassium, Week 12, n=58, 90, 87 | 4.17 (0.282) | 4.17 (0.366) | 4.16 (0.352)
  Potassium, Week 24, n=58, 83, 86 | 4.14 (0.326) | 4.17 (0.390) | 4.16 (0.331)
  Potassium, Week 52/WD, n=60, 90, 89 | 4.14 (0.333) | 4.17 (0.363) | 4.16 (0.306)
  Sodium, BL, n=60, 93, 90 | 141.2 (1.53) | 141.3 (1.66) | 140.7 (1.59)
  Sodium, Week 12, n=58, 90, 87 | 141.1 (1.62) | 140.7 (1.81) | 140.8 (1.47)
  Sodium, Week 24, n=58, 83, 86 | 140.9 (1.23) | 141.1 (1.89) | 141.0 (1.69)
  Sodium, Week 52/WD, n=60, 90, 89 | 141.3 (1.42) | 141.6 (1.62) | 141.2 (1.80)
  Urea/BUN, BL, n=60, 93, 90 | 5.0658 (1.50071) | 5.0928 (1.38695) | 4.7116 (1.12591)
  Urea/BUN, Week 12, n=58, 90, 87 | 5.0792 (1.18333) | 4.9865 (1.23302) | 4.7973 (1.37172)
  Urea/BUN, Week 24, n=58, 83, 86 | 5.0177 (1.16880) | 4.9593 (1.23301) | 4.8510 (1.24616)
  Urea/BUN, Week 52/WD, n=60, 90, 89 | 4.9932 (1.28828) | 4.9869 (1.41120) | 4.7120 (1.16694)

11. Secondary Outcome: Laboratory Parameter of Urine Potential of Hydrogen (pH) at Baseline (Week -2), Week 12, Week 24, and Week 52/WD
Description: Urine samples were collected for measurement at the following scheduled time points: Baseline (Week -2), Week 12, Week 24 and Week 52/WD.
Time Frame: Baseline (Week -2), Week 12, Week 24, and Week 52/WD
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Number analyzed (Participants) | 60 | 93 | 90
pH
  Urine pH, Baseline, n=60, 93, 90 | 6.33 (0.774) | 6.36 (0.883) | 6.46 (0.852)
  Urine pH, Week 12, n=58, 90, 87 | 6.41 (0.726) | 6.36 (0.798) | 6.39 (0.833)
  Urine pH, Week 24, n=58, 83, 86 | 6.27 (0.785) | 6.40 (0.878) | 6.33 (0.807)
  Urine pH, Week 52/WD, n=60, 90, 89 | 6.25 (0.795) | 6.50 (0.775) | 6.42 (0.847)

12. Secondary Outcome: Laboratory Parameter of Urine Specific Gravity (USG) at Baseline (Week -2), Week 12, Week 24, and Week 52/WD
Description: as for outcome 11
Time Frame: Baseline (Week -2), Week 12, Week 24, and Week 52/WD
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio of urine density to water density
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Number analyzed (Participants) | 60 | 93 | 90
ratio of urine density to water density
  Urine Specific Gravity, Baseline, n=60, 93, 90 | 1.0177 (0.00764) | 1.0177 (0.00830) | 1.0173 (0.00734)
  Urine Specific Gravity, Week 12, n=58, 90, 87 | 1.0171 (0.00731) | 1.0167 (0.00789) | 1.0163 (0.00806)
  Urine Specific Gravity, Week 24, n=58, 83, 86 | 1.0174 (0.00795) | 1.0180 (0.00755) | 1.0179 (0.00758)
  Urine Specific Gravity, Week 52/WD, n=60, 90, 89 | 1.0160 (0.00689) | 1.0159 (0.00755) | 1.0156 (0.00811)

13. Secondary Outcome: Number of Participants for the Indicated Uninalysis Parameters Tested by Dipstick at Baseline (BL), Week 12, Week 24, and Week 52/WD
Description: Urinalysis parameters included: Urine Occult Blood (UOB), Urine Glucose (UG), Urine Ketones (UK), Urine Protein (UP), and Urine Leukocyte Esterase test for detecting White Blood Cell (UWBC). The dipstick was a strip used to detect the presence or absence of these parameters in the urine sample. The dipstick test gives results in a semi-quantitative manner, and results can be read as negative (Neg), Trace (TRA), 1+, 2+, and 3+, indicating proportional concentrations in the urine sample. Data are reported as the number of participants who had neg, trace, 1+, 2+, and 3+ levels at Baseline (Week -2) and Week 52/WD.
Time Frame: Baseline (Week -2), Week 12, Week 24, and Week 52/WD
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Number analyzed (Participants) | 60 | 93 | 90
Participants
  UOB, Neg, BL, n=60, 93, 90 | 51 | 79 | 81
  UOB, TRA, BL, n=60, 93, 90 | 6 | 5 | 2
  UOB, 1+, BL, n=60, 93, 90 | 2 | 5 | 2
  UOB, 2+, BL, n=60, 93, 90 | 1 | 3 | 3
  UOB, 3+, BL, n=60, 93, 90 | 0 | 1 | 2
  UOB, Neg, Week 12, n=58, 90, 87 | 50 | 79 | 75
  UOB, TRA, Week 12, n=58, 90, 87 | 2 | 4 | 5
  UOB, 1+, Week 12, n=58, 90, 87 | 4 | 2 | 3
  UOB, 2+, Week 12, n=58, 90, 87 | 2 | 3 | 1
  UOB, 3+, Week 12, n=58, 90, 87 | 0 | 2 | 3
  UOB, Neg, Week 24, n=58, 83, 86 | 49 | 71 | 78
  UOB, TRA, Week 24, n=58, 83, 86 | 4 | 6 | 2
  UOB, 1+, Week 24, n=58, 83, 86 | 1 | 1 | 4
  UOB, 2+, Week 24, n=58, 83, 86 | 3 | 3 | 0
  UOB, 3+, Week 24, n=58, 83, 86 | 1 | 2 | 2
  UOB, Neg, Week 52/WD, n=60, 90, 89 | 54 | 76 | 81
  UOB, TRA, Week 52/WD, n=60, 90, 89 | 4 | 4 | 2
  UOB, 1+, Week 52/WD, n=60, 90, 89 | 0 | 6 | 1
  UOB, 2+, Week 52/WD, n=60, 90, 89 | 1 | 3 | 3
  UOB, 3+, Week 52/WD, n=60, 90, 89 | 1 | 1 | 2
  UG, Neg, BL, n=60, 93, 90 | 58 | 93 | 87
  UG, TRA, BL, n=60, 93, 90 | 2 | 0 | 1
  UG, 1+, BL, n=60, 93, 90 | 0 | 0 | 0
  UG, 2+, BL, n=60, 93, 90 | 0 | 0 | 2
  UG, 3+, BL, n=60, 93, 90 | 0 | 0 | 0
  UG, Neg, Week 12, n=58, 90, 87 | 55 | 90 | 83
  UG, TRA, Week 12, n=58, 90, 87 | 2 | 0 | 0
  UG, 1+, Week 12, n=58, 90, 87 | 1 | 0 | 0
  UG, 2+, Week 12, n=58, 90, 87 | 0 | 0 | 1
  UG, 3+, Week 12, n=58, 90, 87 | 0 | 0 | 3
  UG, Neg, Week 24, n=58, 83, 86 | 53 | 80 | 82
  UG, TRA, Week 24, n=58, 83, 86 | 2 | 1 | 0
  UG, 1+, Week 24, n=58, 83, 86 | 2 | 1 | 1
  UG, 2+, Week 24, n=58, 83, 86 | 1 | 0 | 0
  UG, 3+, Week 24, n=58, 83, 86 | 0 | 1 | 3
  UG, Neg, Week 52/WD, n=60, 90, 89 | 59 | 87 | 84
  UG, TRA, Week 52/WD, n=60, 90, 89 | 0 | 3 | 3
  UG, 1+, Week 52/WD, n=60, 90, 89 | 1 | 0 | 0
  UG, 2+, Week 52/WD, n=60, 90, 89 | 0 | 0 | 1
  UG, 3+, Week 52/WD, n=60, 90, 89 | 0 | 0 | 1
  UK, Neg, BL, n=60, 93, 90 | 60 | 93 | 90
  UK, TRA, BL, n=60, 93, 90 | 0 | 0 | 0
  UK, 1+, BL, n=60, 93, 90 | 0 | 0 | 0
  UK, 2+, BL, n=60, 93, 90 | 0 | 0 | 0
  UK, 3+, BL, n=60, 93, 90 | 0 | 0 | 0
  UK, Neg, Week 12, n=58, 90, 87 | 58 | 89 | 86
  UK, TRA, Week 12, n=58, 90, 87 | 0 | 0 | 0
  UK, 1+, Week 12, n=58, 90, 87 | 0 | 1 | 1
  UK, 2+, Week 12, n=58, 90, 87 | 0 | 0 | 0
  UK, 3+, Week 12, n=58, 90, 87 | 0 | 0 | 0
  UK, Neg, Week 24, n=58, 83, 86 | 58 | 83 | 86
  UK, TRA, Week 24, n=58, 83, 86 | 0 | 0 | 0
  UK, 1+, Week 24, n=58, 83, 86 | 0 | 0 | 0
  UK, 2+, Week 24, n=58, 83, 86 | 0 | 0 | 0
  UK, 3+, Week 24, n=58, 83, 86 | 0 | 0 | 0
  UK, Neg, Week 52/WD, n=60, 90, 89 | 59 | 90 | 89
  UK, TRA, Week 52/WD, n=60, 90, 89 | 0 | 0 | 0
  UK, 1+, Week 52/WD, n=60, 90, 89 | 1 | 0 | 0
  UK, 2+, Week 52/WD, n=60, 90, 89 | 0 | 0 | 0
  UK, 3+, Week 52/WD, n=60, 90, 89 | 0 | 0 | 0
  UP, Neg, BL, n=60, 93, 90 | 55 | 76 | 79
  UP, TRA, BL, n=60, 93, 90 | 4 | 16 | 9
  UP, 1+, BL, n=60, 93, 90 | 1 | 1 | 2
  UP, 2+, BL, n=60, 93, 90 | 0 | 0 | 0
  UP, 3+, BL, n=60, 93, 90 | 0 | 0 | 0
  UP, Neg, Week 12, n=58, 90, 87 | 52 | 82 | 76
  UP, TRA, Week 12, n=58, 90, 87 | 5 | 5 | 7
  UP, 1+, Week 12, n=58, 90, 87 | 0 | 2 | 4
  UP, 2+, Week 12, n=58, 90, 87 | 1 | 0 | 0
  UP, 3+, Week 12, n=58, 90, 87 | 0 | 1 | 0
  UP, Neg, Week 24, n=58, 83, 86 | 50 | 73 | 80
  UP, TRA, Week 24, n=58, 83, 86 | 7 | 8 | 5
  UP, 1+, Week 24, n=58, 83, 86 | 1 | 1 | 1
  UP, 2+, Week 24, n=58, 83, 86 | 0 | 1 | 0
  UP, 3+, Week 24, n=58, 83, 86 | 0 | 0 | 0
  UP, Neg, Week 52/WD, n=60, 90, 89 | 54 | 70 | 68
  UP, TRA, Week 52/WD, n=60, 90, 89 | 5 | 15 | 17
  UP, 1+, Week 52/WD, n=60, 90, 89 | 1 | 4 | 2
  UP, 2+, Week 52/WD, n=60, 90, 89 | 0 | 1 | 2
  UP, 3+, Week 52/WD, n=60, 90, 89 | 0 | 0 | 0
  UWBC, Neg, BL, n=60, 93, 90 | 53 | 79 | 82
  UWBC,TRA, BL, n=60, 93, 90 | 0 | 0 | 0
  UWBC,1+, BL, n=60, 93, 90 | 3 | 7 | 3
  UWBC,2+, BL, n=60, 93, 90 | 3 | 3 | 2
  UWBC,3+, BL, n=60, 93, 90 | 1 | 4 | 3
  UWBC,Neg, Week 12, n=58, 90, 87 | 52 | 73 | 77
  UWBC,TRA, Week 12, n=58, 90, 87 | 0 | 0 | 0
  UWBC,1+, Week 12, n=58, 90, 87 | 2 | 5 | 7
  UWBC,2+, Week 12, n=58, 90, 87 | 3 | 5 | 3
  UWBC,3+, Week 12, n=58, 90, 87 | 1 | 7 | 0
  UWBC,Neg, Week 24, n=58, 83, 86 | 50 | 70 | 78
  UWBC,TRA, Week 24, n=58, 83, 86 | 0 | 0 | 0
  UWBC,1+, Week 24, n=58, 83, 86 | 4 | 6 | 7
  UWBC,2+, Week 24, n=58, 83, 86 | 2 | 5 | 1
  UWBC,3+, Week 24, n=58, 83, 86 | 2 | 2 | 0
  UWBC,Neg, Week 52/WD, n=60, 90, 89 | 52 | 75 | 78
  UWBC,TRA, Week 52/WD, n=60, 90, 89 | 0 | 0 | 0
  UWBC,1+, Week 52/WD, n=60, 90, 89 | 4 | 6 | 2
  UWBC,2+, Week 52/WD, n=60, 90, 89 | 3 | 5 | 7
  UWBC,3+, Week 52/WD, n=60, 90, 89 | 1 | 4 | 2

14. Secondary Outcome: Change From Baseline in the 24-hour Urinary Cortisol Excretion
Description: Urine samples were collected for measurement of urinary cortisol excretion at the following scheduled time points: Baseline (Week 0), Week 24, and Week 52/WD. The 24-hour urinary cortisol excretion was calculated by multiplying the total volume of urine by the concentration of urinary cortisol. Cortisol is a hormone released from the adrenal gland that helps in fat, protein, and carbohydrate metabolism. Change from Baseline was calculated as the value at post-Baseline time point minus the value at Baseline.
Time Frame: Baseline (Week 0), Week 24, and Week 52/WD
Population: Urine cortisol (UC) Population: all participants in the ITT Population from whom urine specimens were collected and who were considered not to have any confounding factors that might affect the analysis of the results of the specimens. Only those participants with post-Baseline data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles (nmol)/24 hours
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Number analyzed (Participants) | 19 | 20 | 28
Nanomoles (nmol)/24 hours
  Week 24, n=19, 20, 28 | 1.0218 (42.309) | 1.0602 (64.825) | 0.9698 (67.211)
  Week 52/WD, n=18, 19, 30 | 0.8956 (48.231) | 1.0802 (73.912) | 0.8190 (41.301)

15. Secondary Outcome: Change From Baseline in Blood Pressure
Description: Blood pressure measurement included systolic blood pressure (SBP) and diastolic blood pressure (DBP) at Baseline (Week 0), Weeks 12, 24 and Week 52/WD. Blood pressure was measured in a sitting position after a participant was kept at rest for at least 5 minutes. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Week 0), Week 12, Week 24, and Week 52/WD
Population: ITT Population. Only those participants with post-Baseline data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Number analyzed (Participants) | 60 | 92 | 89
Millimeters of Mercury (mmHg)
  SBP, Week 12, n=58, 90, 88 | -1.6 (9.54) | 1.2 (11.42) | 0.7 (13.01)
  SBP, Week 24, n=58, 83, 86 | -0.7 (11.76) | -1.6 (12.88) | 0.1 (9.39)
  SBP Week 52/WD, n=60, 92, 89 | -1.5 (9.34) | 0.5 (11.95) | 0.9 (11.66)
  DBP, Week 12, n=58, 90, 88 | -0.3 (8.09) | 1.0 (8.63) | -2.3 (9.28)
  DBP, Week 24, n=58, 83, 86 | -0.7 (8.46) | 0.5 (9.43) | -1.1 (7.82)
  DBP, Week 52/WD, n=60, 92, 89 | -0.1 (8.55) | 1.5 (10.13) | -0.1 (9.20)

16. Secondary Outcome: Change From Baseline in Heart Rate (HR)
Description: Heart rate was measured in a sitting position after a participant was kept at rest for at least 5 minutes at Baseline (Week 0), Weeks 12, 24 and Week 52/WD. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Week 0), Week 12, Week 24, and Week 52/WD
Population: ITT Population. Only those participants with post-Baseline data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats/Minute
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Number analyzed (Participants) | 60 | 92 | 89
Beats/Minute
  Week 12, n=58, 90, 88 | 0.9 (12.27) | -0.6 (9.02) | 1.3 (8.54)
  Week 24, n=58, 83, 86 | 0.1 (9.24) | 0.1 (9.18) | 1.1 (9.97)
  Week 52/WD, n=60, 92, 89 | -1.2 (10.91) | -1.4 (9.62) | 1.1 (9.10)

17. Secondary Outcome: Number of Participants With Abnormal 12-lead Electrocardiogram (ECG) Findings
Description: A 12-lead ECG was recorded in a supine position after the participant was kept at rest in this position for at least 5 minutes at assessment time points (Baseline[Week -2], Week 12, 24 and Week 52/WD) in the treatment period. Data are presented for clinically significant (CS) as well as not clinically significant (NCS) abnormal (Abn) findings. Any abnormal ECG, including those that worsen from Baseline, and determined clinically significant by the assessment of the investigator were recorded as CS.
Time Frame: Week 12, Week 24, and Week 52/WD
Population: ITT Population. . Only participants remaining in the study and contributing evaluable data at the indicated time points were analyzed.; thus the number of participants analyzed reflects everyone in the ITT Population. The number of participants assessed for each parameter is indicated by "n=X, X".
Measure: Number; unit: Participants
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Number analyzed (Participants) | 60 | 93 | 90
Participants
  Baseline, Abn NCS, n=60, 93, 90 | 19 | 22 | 11
  Baseline, Abn CS, n=60, 93, 90 | 0 | 0 | 0
  Week 12, Abn NCS, n=58, 90, 88 | 11 | 17 | 10
  Week 12, Abn CS, n=58, 90, 88 | 0 | 0 | 0
  Week 24, Abn NCS, n=58, 83, 86 | 12 | 18 | 9
  Week 24, Abn CS, n=58, 83, 86 | 0 | 0 | 0
  Week 52/WD, Abn NCS, n=60, 90, 89 | 10 | 16 | 12
  Week 52/WD, Abn CS, n=60, 90, 89 | 0 | 2 | 0

18. Secondary Outcome: Number of Participants With Severe Asthma Exacerbation During the Study Treatment
Description: A severe asthma exacerbation is defined as the deterioration of asthma requiring the use of systemic corticosteroids (tablets, suspension, or injection) for at least 3 days or an in-patient hospitalization or emergency department visit due to asthma that required systemic corticosteroids. Courses of corticosteroids separated by 1 week or more were treated as separate severe exacerbations.
Time Frame: Baseline up to Week 52
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Number analyzed (Participants) | 60 | 93 | 90
Participants | 3 | 9 | 16

19. Secondary Outcome: Change From Baseline in Diary Data - Morning (AM) Peak Expiratory Flow (PEF) and Evening (PM) PEF During the Study Treatment
Description: Change from Baseline in AM and PM PEF at 52 weeks of evaluation period during study treatment was recorded in the dairy record card. The Baseline value was calculated as the mean of all available data recorded during the7 days immediately prior to the treatment start date (including Day 1: Day 1 is treatment start date). The PEF is defined as the greatest rate of airflow that can be achieved during forced exhalation beginning with the lungs fully inflated.
Time Frame: Baseline up to Week 52
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Litres per Minute (L/min)
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Number analyzed (Participants) | 60 | 93 | 90
Litres per Minute (L/min)
  PEF AM, Week 0-52 | 18.29 (36.304) | 23.98 (38.668) | 12.38 (32.295)
  PEF PM, Week 0-52 | 20.23 (35.274) | 26.29 (40.510) | 15.64 (30.772)

20. Secondary Outcome: Change From Baseline in Asthma Symptom Score During the Study Treatment
Description: The Baseline value was calculated as the mean of all available data recorded during the 7 days immediately prior to Visit 2 (treatment assignment visit). Participants entered their asthma symptom score in the patient diary twice daily (morning and evening). Daytime asthma symptom scores: 0-no asthma symptoms, 1-one episode of short-time asthma symptoms, 2-two or more episodes of short-time asthma symptoms, 3-asthma symptoms occurring during most part of daytime without interference with daily life activities, 4-asthma symptoms occurring during most part of daytime with interference with daily life activities, 5-severe asthma symptoms that disable working or daily life activities. Nighttime asthma symptom scores: 0-no asthma symptoms, 1-one awakening due to asthma symptoms, 2-two or more awakenings due to asthma symptoms, 3-asthma symptoms almost prevented the participant from sleeping, 4-severe asthma symptoms completely prevented from sleeping.
Time Frame: Baseline up to Week 52
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Number analyzed (Participants) | 60 | 93 | 90
Scores on a scale | -0.14 (0.638) | -0.14 (0.856) | -0.19 (0.771)

21. Secondary Outcome: Change From Baseline in the Percentage of Symptom-free 24-hour Periods During the Study Treatment
Description: Participants who were symptom free for 24-hours were assessed. Change from Baseline is calculated as the value at Week 52 minus the value at Baseline.
Time Frame: Baseline up to Week 52
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Percentage of symptom-free days
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Number analyzed (Participants) | 60 | 93 | 90
Percentage of symptom-free days | 6.79 (20.382) | 6.51 (28.290) | 8.19 (26.975)

22. Secondary Outcome: Change From Baseline in the Percentage of Rescue-free 24-hour Periods
Description: The time span during which the participants did not have to take any rescue medication (medication intended to relieve symptoms immediately) was considered as a rescue free period. Change from Baseline is calculated as the value at Week 52 minus the value at Baseline.
Time Frame: Baseline up to Week 52
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Percentage of rescue free 24-hour period
Groups:
- FF 100 µg: Participants received FF/GW642444 inhalation powder 200/25 µg OD in the evening from the DPI over the 52 week treatment period.
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Number analyzed (Participants) | 60 | 93 | 90
Percentage of rescue free 24-hour period
  Week 0-12, n=60, 93, 90 | 97.94 (9.553) | 95.51 (16.427) | 92.79 (17.462)
  Week 13-24, n=58, 91, 88 | 97.60 (7.521) | 95.94 (13.477) | 94.35 (16.990)
  Week 25-36, n=58, 84, 87 | 97.99 (8.757) | 95.24 (14.685) | 94.14 (15.713)
  Week 37-52, n=57, 79, 86 | 98.38 (7.253) | 95.71 (13.382) | 95.13 (14.705)
  Week 0-52, n=60, 93, 90 | 98.01 (7.736) | 95.76 (13.556) | 94.28 (15.169)

23. Secondary Outcome: Number of Rescue Medication Inhalations
Description: Salbutamol inhaler was used as the rescue medication. Participants entered the number of rescue medication inhalations in the patient diary twice daily (morning and evening).
Time Frame: Baseline up to Week 52
Population: ITT Population. The number of participants analyzed depends on the number of participants remaining in the indaicated time period.
Measure: Mean (Standard Deviation); unit: Number of inhalations
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Number analyzed (Participants) | 60 | 93 | 90
Number of inhalations
  Week 0-12, n=60, 93, 90 | 5.15 (31.288) | 7.32 (27.667) | 13.42 (43.889)
  Week 13-24, n=58, 91, 88 | 5.12 (19.094) | 6.65 (23.257) | 12.56 (54.154)
  Week 25-36, n=58, 84, 87 | 6.02 (36.358) | 7.45 (25.058) | 14.01 (70.642)
  Week 37-52, n=57, 79, 86 | 7.75 (50.851) | 7.73 (22.285) | 17.78 (97.092)
  Week 0-52, n=60, 93, 90 | 23.28 (132.467) | 27.13 (90.038) | 56.23 (253.508)

ADVERSE EVENTS:
Time Frame: On-treatment non-serious adverse events (AEs), defined as those events occurring while participants were on treatment, up to and including the day after the last dose in each treatment period (up to 52 weeks), are reported. SAEs, defined as those events o
Description: SAEs and non-serious AEs were collected in the Intent-to-Treat (ITT) Population, comprised of all participants randomized to treatment who received at least one dose of study medication.
Arm/Group | FF/GW642444 100/25 µg | FF/GW642444 200/25 µg | FF 100 µg
Serious Adverse Events (participants affected / at risk) | 4/60 | 7/93 | 1/90
Other Adverse Events (participants affected / at risk) | 52/60 | 77/93 | 72/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FF/GW642444 100/25 µg (N=60) | FF/GW642444 200/25 µg (N=93) | FF 100 µg (N=90)
Pneumonia (Infections and infestations) | 1 | 1 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis hypertrophic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FF/GW642444 100/25 µg (N=60) | FF/GW642444 200/25 µg (N=93) | FF 100 µg (N=90)
Nasopharyngitis (Infections and infestations) | 37 | 57 | 49
Bronchitis (Infections and infestations) | 8 | 18 | 12
Pharyngitis (Infections and infestations) | 7 | 12 | 12
Oral candidiasis (Infections and infestations) | 3 | 13 | 3
Influenza (Infections and infestations) | 2 | 9 | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 6
Gastroenteritis (Infections and infestations) | 7 | 0 | 7
Headache (Nervous system disorders) | 5 | 4 | 5
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 6 | 1
Eczema (Skin and subcutaneous tissue disorders) | 4 | 3 | 3
Abdominal discomfort (Gastrointestinal disorders) | 3 | 0 | 4
Alanine aminotransferase increased (Investigations) | 3 | 2 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4 | 0 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2
Conjunctivitis allergic (Eye disorders) | 3 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 5
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.